CLINICAL TRIAL: NCT04136275
Title: A Phase I Clinical Trial with CAR-37 T Cells for the Treatment of Patients with Relapsed or Refractory CD37+ Hematologic Malignancies
Brief Title: CAR-37 T Cells in Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Marcela V. Maus, M.D.,Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Marcela V. Maus, M.D.,Ph.D., Sponsor Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-087
Record Dates: First submitted 2019-10-19; First posted 2019-10-23 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Hematologic Malignancy; Leukemia; Lymphoma; Lymphoma, B-Cell; Lymphoma, T-Cell; Lymphoma, Non-Hodgkin
Keywords: Leukemia; Hematologic Malignancy; Lymphoma; CAR-T
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Lymphoma, B-Cell; Lymphoma, T-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAR-37 T cells (Experimental): * CAR-37 will be administered intravenously on day 0
  * Enrolled subjects will undergo a leukapheresis procedure processing approximately two times the subject's total blood volume.
  * Subjects will receive 3 days of lymphodepleting chemotherapy starting Day -5, before the infusion of CAR-37 T cells on Day 0
  Interventions: Biological: CAR-37 T cells
- CAR-37 T cells Dose Escalation (Experimental): * CAR-37 will be administered intravenously on day 0
  * Enrolled subjects will undergo a leukapheresis procedure processing approximately two times the subject's total blood volume.
  * CAR-37 will undergo dose escalation
  Interventions: Biological: CAR-37 T cells

INTERVENTIONS:
Biological: CAR-37 T cells — CAR-37 is an investigational treatment that uses the participant own immune cells, called T cells, to try to kill the cancerous cells

SUMMARY:
This research study is studying Chimeric Antigen Receptor (CAR)-37 T Cells (CAR-37 T Cells) for treating people with relapsed or refractory CD37+ hematologic malignancies and to understand the side effects when treated with CAR-37 T Cells.

- Chimeric Antigen Receptor (CAR)-37 T Cells (CAR-37 T Cells) is an investigational treatment

DETAILED DESCRIPTION:
This is a two-part, non randomized, open label, single site Phase 1 study. Participants who fulfill eligibility criteria will be entered into the trial Chimeric Antigen Receptor (CAR)-37 T Cells (CAR-37 T Cells).

This study consists of 2 parts:

* Part A (Dose Escalation): The investigators are looking the highest dose of the study intervention that can be administered safely without severe or unmanageable side effects in participants that have relapsed or refractory CD37+ hematologic malignancies, not everyone who participates in this research study will receive the same dose of the study intervention. The dose given will depend on the number of participants who have been enrolled prior and how well the dose was tolerated
* Part B (Expansion Cohort): Part B: Expansion Cohort: Participants will be treated at the respective dose (at or below the Maximum Tolerated Dose), as determined during Part A (Dose Escalation).
* A total of 18 participants will be enrolled to this trial

This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies.

Investigational" means that the intervention is being studied The U.S. Food and Drug Administration (FDA) has not approved CAR-37 T Cells as a treatment for any disease.

This is the first time that CAR-37 T Cells will be given to humans

ELIGIBILITY:
Inclusion Criteria:

Voluntarily sign informed consent form.

Age ≥18 years of at the time of signing informed consent

Eastern Cooperative Oncology Group (ECOG) performance status 0-2 Karnofsky ≥60%, see Appendix A)

* Diagnosis of relapsed/refractory (R/R) CD37+ hematologic malignancy as defined as one of the following:
* Mature B cell neoplasms

  * Follicular Lymphoma (FL) grade 1, grade 2, or grade 3a

    * RR disease after 2 or more prior lines of therapy AND
    * 1 of the prior lines of therapy must include an anti-CD20 antibody monotherapy.
  * Marginal Zone Lymphoma (MZL) nodal or extranodal:

    * R/R disease after 2 or more prior lines of therapy AND
    * 1 of the prior lines of therapy must include an anti-CD20 antibody monotherapy
  * Diffuse large B-cell lymphoma (DLBCL), including transformed follicular lymphoma (FL), primary mediastinal B-cell lymphoma (PMBCL), high-grade B-cell lymphoma and grade 3b Follicular Lymphoma (FL).

    * R/R disease after 2 or more prior lines of therapy OR
    * Relapsed following autologous SCT,OR
    * Ineligible for autologous SCT.
  * Mantle cell lymphoma

    * R/R disease as defined by disease progression after last regimen (including autologous SCT), OR Refractory disease as defined as failure to achieve a CR to last regimen.
    * Prior therapy must include:

      * Anthracycline or bendamustine-containing chemotherapy AND
      * Anti-CD20 monoclonal antibody therapy AND
      * BTKi therapy
  * Chronic lymphocytic leukemia (CLL)

    * CLL with an indication for treatment based on iwCLL guidelines and clinical measurable disease (lymphocytosis > 5×109/L and/or measurable lymph nodes and/or hepatic or splenomegaly)
    * Subjects must have received previous treatment as follows:

      * Subjects with high-risk features, defined as having complex cytogenetic abnormalities (3 or more chromosomal abnormalities), 17p deletion, TP53 mutation, or unmutated IGHV, must have failed at least 1 line of prior therapy, including a BTKi OR
      * Subjects with standard-risk features must have failed at least 2 lines of prior therapy, including a BTKi OR
      * Subjects who are BTKi intolerant and have received < 6 months of BTKi therapy, must have failed at least 1 high-risk line of non-BTKi therapy or 2 standard-risk lines of non-BTKi therapy OR
      * Subjects who are ineligible for BTKi, must have failed at least 1 (high-risk) line of non-BTKi therapy or 2 (standard-risk) lines of non-BTKi therapy.
  * Small lymphocytic lymphoma (SLL)

    * SLL (lymphadenopathy) or SLL (splenomegaly and < 5x 109 CD19+ CD5+ clonal B lymphocytes/L [<5000/μL] in the peripheral blood at diagnosis with measurable disease defined as at least one lesion > 1/5 cm in the greatest transverse diameter that is biopsy-proven SLL)
    * Subjects must have received previous treatments as follows:

      * Subjects with high-risk features, defined as having complex cytogenetic abnormalities (3 or more chromosomal abnormalities), or 17p deletion, or TP53 mutation, or unmutated IGHV, must have failed at least 1 line of prior therapy, including a BTKi OR
      * Subjects with standard-risk features must have failed at least 2 lines of prior therapy, including a BTKi OR
      * Subjects who are BTKi intolerant and have received < 6 months of BTKi therapy must have failed at least 1 high-risk or 2 standard-risk other lines of non-BTKi therapy OR
      * Subjects who are ineligible for BTKi, must have failed at least 1 high-risk or 2 standard-risk other lines of non-BTKi therapy.
  * Mature T cell neoplasms:

    * Peripheral T-Cell lymphoma (PTCL)/Cutaneous T-Cell Lymphoma (CTCL)
    * R/R after 2 or more prior lines of therapy OR
    * Relapse following autologous stem cell transplant OR
  * T-cell prolymphocytic leukemia (TPLL) --- Diagnosis of TPLL with plan for subsequent therapy.
* Evidence of CD37 expression on tumor cells as demonstrated by flow cytometry and/or IHC on fresh biopsy or historic samples.
* Subjects must have measurable disease according to appropriate disease specific criteria.
* Adequate absolute lymphocyte count (ALC > 100 cells/ul) within one week of apheresis.
* Adequate bone marrow function defined by absolute neutrophil count (ANC) >1000 cells/mm3 without growth factor support (filgrastim within 7 days of pegfilgrastim within 14 days) and untransfused platelet count >50,000 mm3.
* Left ventricular ejection fraction > 40%
* Adequate hepatic function defined by aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) < 2.5 × upper limit of normal (ULN) and direct bilirubin < 1.5 × ULN.
* Adequate renal function defined by creatinine clearance >30 ml/min using the Cockcroft-Gault formula.
* The effects of CAR-37 T cells on the developing human fetus are unknown. For this reason, women of child-bearing potential and men with partners of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to leukapheresis and until 6 months post CAR-37 infusion. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men with partners of childbearing potential treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and until 4 months after last CAR-37 T cells administration.
* Ability and willingness to adhere to the study visit schedule and all protocol requirements

Inclusion criteria for lymphodepletion:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Karnofsky ≥60%, see Appendix A).
* No Active, uncontrolled, systemic bacterial, viral, or fungal infection. If febrile, the patient must be afebrile for 24 hours and blood cultures negative for 48 hours on appropriate antibiotic therapy.
* Oxygen saturation >92% on room air while awake.
* No additional anti-cancer therapy since leukapheresis excluding steroids at or below physiologic dosing.

Exclusion Criteria:

* Prior CD37 targeted therapies.
* Treatment with an any investigational cellular therapy within 8 weeks prior to apheresis.
* Any systemic anti-cancer therapy within 1 weeks of leukapheresis excluding steroids at or below physiologic dosing.
* Ongoing treatment with chronic immunosuppressants (e.g., cyclosporine or systemic steroids above physiologic dosing). Intermittent topical, inhaled, or intranasal corticosteroids are allowed.
* Ongoing systemic immunosuppression for acute and/or chronic GVH as a result of previous allogeneic bone marrow transplant and at least 12 weeks out from prior allogeneic SCT.
* Significant co-morbid condition or disease which in the judgment of the Principal Investigator would place the subject at undue risk or interfere with the study; examples include, but are not limited to, cirrhotic liver disease, sepsis, and/or recent significant traumatic injury.
* Active, uncontrolled, systemic bacterial, viral, or fungal infection.
* Subjects with a history of class III or IV congestive heart failure or with a history of non- ischemic cardiomyopathy.
* Subjects with unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the previous 3 months.
* Subjects with arterial vascular disease such as history of cerebrovascular accident or peripheral vascular disease requiring therapeutic anti-coagulation.
* Subjects with history of a new pulmonary embolism within 6 months of beginning lymphodepletion.
* Subjects with second malignancies if the second malignancy has required therapy in the last 3 years or is not in complete remission; exceptions to this criterion include successfully treated non-metastatic basal cell or squamous cell skin carcinoma, or prostate cancer that does not require therapy other than hormonal therapy.
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 2 years
The occurrence of study related adverse events | 2 years

SECONDARY OUTCOMES:
Disease Specific Response | 2 years
Overall Survival | 2 years
Progression Free Survival | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Frigault, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to the Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Background] Scarfo I, Ormhoj M, Frigault MJ, Castano AP, Lorrey S, Bouffard AA, van Scoyk A, Rodig SJ, Shay AJ, Aster JC, Preffer FI, Weinstock DM, Maus MV. Anti-CD37 chimeric antigen receptor T cells are active against B- and T-cell lymphomas. Blood. 2018 Oct 4;132(14):1495-1506. doi: 10.1182/blood-2018-04-842708. Epub 2018 Aug 8. PMID 30089630
- [Derived] Frigault MJ, Graham CE, Berger TR, Ritchey J, Horick NK, El-Jawahri A, Scarfo I, Schmidts A, Haradhvala NJ, Wehrli M, Lee WH, Parker AL, Wiggin HR, Bouffard A, Dey A, Leick MB, Katsis K, Elder EL, Dolaher MA, Cook DT, Chekmasova AA, Huang L, Nikiforow S, Daley H, Ritz J, Armant M, Preffer F, DiPersio JF, Nardi V, Chen YB, Gallagher KME, Maus MV. Phase 1 study of CAR-37 T cells in patients with relapsed or refractory CD37+ lymphoid malignancies. Blood. 2024 Sep 12;144(11):1153-1167. doi: 10.1182/blood.2024024104. PMID 38781564